CLINICAL TRIAL: NCT05917678
Title: Effectiveness of Repositioning, Physical Therapy, and Cranial Remolding in Infants With Cranial Deformation
Brief Title: Effectiveness of Repositioning and Cranial Remolding in Infants With Cranial Deformation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Children's Health (Other)
Responsible Party: Principal Investigator, Tiffany Graham, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 032017-036
Record Dates: First submitted 2023-06-05; First posted 2023-06-26 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Deformational Plagiocephaly; Deformational Posterior Plagiocephaly; Brachycephaly; Torticollis; Congenital Muscular Torticollis
Keywords: plagiocephaly; brachycephaly; asymmetrical brachycephaly; helmet; cranial remolding; orthosis; repositioning; deformational; torticollis; normal
MeSH Terms: conditions — Plagiocephaly, Nonsynostotic; Craniosynostoses; Torticollis; Congenital torticollis; Plagiocephaly | interventions — Head Protective Devices

STUDY DESIGN:
Intervention Model Description: Infants with deformational head shapes start with repositioning strategies, then some will change to the orthotic intervention (custom remolding helmet). Healthy infants will only be followed, no intervention performed. All infants will be followed until 12 months of age.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Repositioning Therapy (Other): Infants will be treated with at-home repositioning strategies for their deformational head shape. Physical therapy will be provided, if indicated, for treatment of torticollis. This is a standard treatment.
  Interventions: Other: Repositioning Therapy
- Repositioning Therapy + Cranial Remolding Orthoses (Other): After attempting at 2-4 months of repositioning therapy, infants with residual cranial deformation may be treated with a custom made helmet (cranial remolding orthosis) which is adjusted every few weeks to direct skull growth. It is worn 23 hours per day. Physical therapy will be provided, if indicated, for treatment of torticollis. This is a standard treatment.
  Interventions: Other: Repositioning Therapy; Device: Cranial Remolding Orthosis
- Control (No Intervention): Healthy infants without deformational head shapes or need for physical therapy will be followed and measured. No intervention.

INTERVENTIONS:
Other: Repositioning Therapy — Caregivers will be instructed how to increase tummy time activities and reshape their infant's heads using at-home methods to direct their attention to the non-preferred side.
  Arms: Repositioning Therapy; Repositioning Therapy + Cranial Remolding Orthoses
Device: Cranial Remolding Orthosis — A custom cranial remolding orthosis (FDA Class II device) will be made to fit affected infants. this should be worn 23 hours per day and the Orthotist needs to be seen regularly for adjustments until the head shape is resolved.
  Other Names: Helmet, Cranial Band, STARband
  Arms: Repositioning Therapy + Cranial Remolding Orthoses

SUMMARY:
This study will examine how effective caregiver's repositioning strategies are in correcting an infant's deformational cranial shape, as well as the effectiveness of the use of a custom cranial remolding orthosis for treatment of deformational head shapes. Infants with torticollis will be concurrently enrolled in physical therapy treatment until the torticollis is resolved. A normal, unaffected population will be studied to compare typical growth to the growth of infants undergoing active treatment.

DETAILED DESCRIPTION:
Infants 2 months of age who have been diagnosed with a deformational head shape will be begin repositioning therapy (and physical therapy if torticollis is present) and be followed at least monthly. At 4, 5, and 6 months of age, if the head shape has not resolved, they will be given the option to pursue treatment with a cranial remolding orthosis. All affected infants will undergo active treatment until the head shape is resolved or the infant is 12 months of age (whichever comes first).

Normal infants will be evaluated at 2, 6, and 12 months of age and will not be enrolled in any active treatment.

All infants will return at 12 months of age for a final evaluation.

ELIGIBILITY:
Inclusion Criteria for Control Group:

* Healthy infants with normal physical development and no need for physical therapy intervention

Exclusion Criteria for Control Group:

* Infants with abnormal head shapes (plagiocephaly or craniosynostosis)
* Infants with growth abnormalities (such as genetic conditions)
* Infants with developmental delay significant to warrant physical therapy or occupational therapy

Ages: 2 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Final Head Shape | 10 months after enrollment (at 12 months of age)
  Cranial measurements will be used to assess residual cranial deformation in affected infants. A group of unaffected, typically-developing infants will be used as normal growth examples.
  Measurements include 2-dimensional measurements (taken at the greater equator of the skull with cranial calipers or a measuring tape): Cranial circumference, medio-lateral dimension of the skull, anterior-posterior dimension of the skull, two opposing diagonal measurements taken 30 degrees from the mid-sagittal line. These will be used to calculate the asymmetry and proportion of the skull and track growth.
  Measurements include 3-dimensional measurements: 1) An FDA-approved non-invasive, eye-safe laser scanner called the STARscanner will be used to track measurements throughout treatment. For those who switch to Cranial Remolding Therapy, this scanner will be used for custom helmet fabrication. 2) The 3dMD system will use photographs to create a 3-dimensional rendering of your child's head.

SECONDARY OUTCOMES:
Overall Change in Head Shape | Assessment to occur within 2 years of enrollment closure.
  The improvements seen in each of the 2 treatment arms will be compared to determine if one treatment has a greater impact than the other treatment.
  Specifically, the difference between the baseline measurements (taken at 2 months of age) and the updated measurements (taken at each study measurement timepoint) will be compared in 2-dimensions and 3-dimensions. The group with greater correction to the cranial deformity would be considered the more impactful treatment method.
Compliance with treatment | Assessment to occur within 2 years of enrollment closure.
  Overall compliance with each treatment method will be assessed.
  Caregivers of affected infants will be given surveys at each follow up appointment to assess adherence to the treatment arm's protocol. Surveys will include questions specific to the infant's treatment arm, which may include questions such as how long the child remains in a repositioned position before moving themselves, how many hours per day the infant is wearing their custom helmet, and how often caregivers are performing the recommended neck stretches.
  No surveys will be given to the typically-developing control group as there is no active treatment for this group.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Graham, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No identifiable data will be shared outside of the study investigators.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT05917678/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT05917678/ICF_001.pdf